CLINICAL TRIAL: NCT02347345
Title: The Immunologic Effects of HCV Therapy With Fixed Dose Combination Ledipasvir/Sofosbuvir (HARVONI) in HCV Genotype 1 Chronically Mono-infected Active and Former IDUs.
Brief Title: Immunologic Effects of HCV Therapy With HARVONI in HCV Genotype 1 Chronically Mono-infected Active and Former IDUs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Martin Markowitz, Aaron Diamond Professor/Clinical Director, Rockefeller University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMA-0874; 5R01DA033777 (NIH)
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C
Keywords: HCV, injection drug use
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active injection drug use (IDU) (Active Comparator): In active IDU, Harvoni (Fixed dose combination ledipasvir/sofosbuvir), one pill orally daily x 12 weeks
  Interventions: Drug: Harvoni (Fixed dose combination ledipasvir/sofosbuvir)
- Former injection drug use (former IDU) (Active Comparator): In former IDU, Harvoni (Fixed dose combination ledipasvir/sofosbuvir), one pill orally daily x 12 weeks
  Interventions: Drug: Harvoni (Fixed dose combination ledipasvir/sofosbuvir)
- Healthy volunteers (No Intervention): HIV, HCV and HBV negative, never injected drugs, no recreational drugs for at least 2 years (does not include marijuana) and negative urine screen for opiates at the screening visit.

INTERVENTIONS:
Drug: Harvoni (Fixed dose combination ledipasvir/sofosbuvir) — Harvoni (Fixed dose combination ledipasvir/sofosbuvir), one pill daily x 12 weeks
  Other Names: Fixed dose combination ledipasvir/sofosbuvir
  Arms: Active injection drug use (IDU); Former injection drug use (former IDU)

SUMMARY:
The investigator's hypothesis is that active injectors will show a partial reduction in markers of immune activation with HCV therapy whereas non-injectors will show a more significant reduction in these markers, and will exhibit levels of immune activation that approach that seen in similarly studied healthy volunteers.This is based on observations that this group of investigators have made. They have shown that individuals who inject drugs have high level of immune activation in blood and tissue. Immune activation or chronic inflammation has been associated with accelerated aging, cardiovascular, renal and liver disease as well as CNS dysfunction. It remains unclear whether increased levels of immune activation are due to non-sterile injection of drugs, chronic infection with Hepatitis C, chronic opiate use, or perhaps combinations of all 3. To understand the potential contribution of infection with Hepatitis C the investigators will compare levels of immune activation pre- and post treatment with an all oral, one pill once daily, interferon sparing treatment of HCV in 2 groups of chronically HCV infected patients- one actively injecting with drugs and the other free of injection for at least 4 months. Immune activation comparisons will also include non-injecting healthy volunteers.

DETAILED DESCRIPTION:
This group of multidisciplinary investigators has discovered increased levels of immune activation among HIV-1-uninfected active injection drug users (IDUs) when compared to non-IDU controls . The vast majority (80%) are also infected with HCV.

Active injectors have high levels of immune activation as measured by sCD14, CD8 co-expression of CD38 and HLA-DR, as well as Type 1 cytokines.

Within months of ceasing injecting, there are observable decreases in some parameters however in general they remain elevated when compared to non-injecting healthy volunteers.

As approximately 80% of these subjects are HCV infected and viremic, these results are confounded as to the cause of the observed increased levels of markers of immune activation- active injection or chronic Hepatitis C. Until recently HCV treatment required the use of IFN which has immunomodulatory activity which would cause perturbations in the markers of immune activation. However the development of direct acting agents (DAA) to treat HCV has revolutionized therapy. In this trial the investigators will employ the once daily FDC formulation of sofosbuvir and ledipasvir to assess changes in markers of immune activation during therapy.

There have been multiple clinical trials of FDC LDV-SOF in patients with Genotype 1 HCV. When taken once daily for 12 weeks, sustained virologic response rates have been very high with response rates nearing 99% in most studies with a 12-week course of therapy.

Common adverse events associated with FDC LDV-SOF in ION-1 include fatigue (21%), headache (25%), nausea (11%), insomnia (8%), asthenia (7%), diarrhea (11%), rash (7%), irritibility (7%), cough (3%), and pruritis (5%).

Ledipasvir undergoes minimal metabolism and expectations are that this medication will have few clinically significant drug-drug interactions. In general, sofosbuvir is considered to have relatively few clinically significant drug-drug interactions, but coadministration of sofosbuvir with the following medications is not recommended because these medications may significantly lower sofosbuvir levels:

Anticonvulsants: carbamazepine, oxycarbazepine, phenobarbital, and phenytoin Antimycobacterials: rifabutin, rifampin, rifapentine Herbal Supplements: St. John's wort HIV Protease Inhibitors: tipranavir-ritonavir Antiarrhythmic Drugs : amiodarone (Cordarone®, Nexterone®, Pacerone®)

Participants will be provided with a 12-week course of FDC LDV-SOF which will provide a near 99% likelihood of a SVR in participants who are adherent to therapy with low likelihood of significant adverse events and drug-drug interactions.

In treating HCV effectively the investigators will measure changes in immune activation and gene expression that accompany HCV treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give written informed consent in English
2. Age≥18 and ≤55
3. HCV antibody positive
4. HCV RNA >1,000 copies/mL plasma
5. HCV treatment naive
6. HCV genotype 1a or 1b or mixed type 1
7. AST, ALT <10x ULN
8. Direct bilirubin <3.0
9. Platelet count >50,000
10. Creatinine clearance >30mL/min as estimated by Cockroft Gault
11. Hemoglobin >10 if female, >11 if male
12. Albumin > 2.8
13. INR<2.0
14. If Group A: urine dip for opiates + and active injection drug use of heroin defined as injecting at least 3 times per week.
15. If Group B then no IDU for at least 4 months and a negative urine for opiates at screening.
16. Venous access for phlebotomy
17. Willingness to agree to effective contraception during the course of the study.
18. If Group C: - negative urine for opiates at screening

    * no recreational drug use for at least 2 years (excluding marijuana)
    * HIV, HCV and HBV uninfected

Exclusion Criteria:

1. HIV infection
2. Chronic infection with Hepatitis B
3. Uncompensated cirrhosis
4. Required use of:

   Anticonvulsants: carbamazepine, oxycarbazepine, phenobarbital, and phenytoin

   Antimycobacterials: rifabutin, rifampin, rifapentine

   Herbal Supplements: St. John's wort

   HIV Protease Inhibitors: tipranavir-ritonavir

   Antiarrhythmic Drugs: amiodarone (Cordarone, Nexterone, Pacerone)
5. Any medical condition that in the opinion of the investigator would interfere with study participation and medical adherence
6. Pregnancy/breast feeding

   -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Markowitz, MD, Principal Investigator — ADARC/Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kowdley KV, Gordon SC, Reddy KR, Rossaro L, Bernstein DE, Lawitz E, Shiffman ML, Schiff E, Ghalib R, Ryan M, Rustgi V, Chojkier M, Herring R, Di Bisceglie AM, Pockros PJ, Subramanian GM, An D, Svarovskaia E, Hyland RH, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Pound D, Fried MW; ION-3 Investigators. Ledipasvir and sofosbuvir for 8 or 12 weeks for chronic HCV without cirrhosis. N Engl J Med. 2014 May 15;370(20):1879-88. doi: 10.1056/NEJMoa1402355. Epub 2014 Apr 10. PMID 24720702
- [Result] Lawitz E, Poordad FF, Pang PS, Hyland RH, Ding X, Mo H, Symonds WT, McHutchison JG, Membreno FE. Sofosbuvir and ledipasvir fixed-dose combination with and without ribavirin in treatment-naive and previously treated patients with genotype 1 hepatitis C virus infection (LONESTAR): an open-label, randomised, phase 2 trial. Lancet. 2014 Feb 8;383(9916):515-23. doi: 10.1016/S0140-6736(13)62121-2. Epub 2013 Nov 5. PMID 24209977
- [Result] Gane EJ, Deray G, Liaw YF, Lim SG, Lai CL, Rasenack J, Wang Y, Papatheodoridis G, Di Bisceglie A, Buti M, Samuel D, Uddin A, Bosset S, Trylesinski A. Telbivudine improves renal function in patients with chronic hepatitis B. Gastroenterology. 2014 Jan;146(1):138-146.e5. doi: 10.1053/j.gastro.2013.09.031. Epub 2013 Sep 22. PMID 24067879

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Injection Drug Use (IDU): In active IDU, Harvoni (Fixed dose combination ledipasvir/sofosbuvir), one pill oral daily x 12 weeks.
- Former Injection Drug Use (Former IDU): In former IDU, Harvoni (Fixed dose combination ledipasvir/sofosbuvir), one pill oral daily x 12 weeks.
- Healthy Volunteers: HIV, HCV, and HBV negative, never injected drugs, no recreational drugs for at least 2 years (does not include marijuana) and negative urine screen for opiates at screening.
Period: Overall Study
Arm/Group | Active Injection Drug Use (IDU) | Former Injection Drug Use (Former IDU) | Healthy Volunteers
Started | 10 | 12 | 12
Completed | 10 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Injection Drug Use (IDU) | Former Injection Drug Use (Former IDU) | Healthy Volunteers | Total
Number analyzed (Participants) | 10 | 12 | 12 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 12 | 34
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 7 | 8 | 8 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 12 | 12 | 34

OUTCOME MEASURES:

1. Primary Outcome: sCD14 (ng/mL)
Description: Marker of immune activation as measured by levels of soluble CD14. Note that the levels of sCD14 were only measured at baseline in the Healthy Volunteers group and therefore there are no data for weeks 4, 12, or 24 entered.
Time Frame: 24 weeks
Population: 9/10 Active injectors, 11/12 former injectors and 12/12 healthy volunteers completed the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Active Injection Drug Use (IDU) | Former Injection Drug Use (Former IDU) | Healthy Volunteers
Number analyzed (Participants) | 10 | 12 | 12
ng/mL
  baseline | 1986 (217) | 1918 (208) | 1542 (249)
  week 4: number analyzed (Participants) | 10 | 12 | 0
  week 4 | 2060 (443) | 1805 (183) |
  week 12: number analyzed (Participants) | 10 | 12 | 0
  week 12 | 2036 (339) | 1782 (193) |
  week 24: number analyzed (Participants) | 9 | 11 | 0
  week 24 | 1973 (266) | 1819 (193) |
Statistical Analysis 1: Comparison: Active Injection Drug Use (IDU) vs Former Injection Drug Use (Former IDU) vs Healthy Volunteers; Test type: Other — Descriptive pilot study. Not relevant; p = 0.07, Kruskal-Wallis

2. Secondary Outcome: Virologic Response to Therapy as Measured by HCV RNA
Description: HCV RNA levels in plasma (IU/mL)
Time Frame: 24 weeks
Population: 9/10 Active injectors, 11/12 former injectors and 12/12 healthy volunteers completed the study. Healthy volunteers are HCV uninfected therefore HCV RNA levels are not measured on this group of participants.
Measure: Mean (Standard Deviation); unit: HCV RNA copies/mL plasma
Arm/Group | Active Injection Drug Use (IDU) | Former Injection Drug Use (Former IDU) | Healthy Volunteers
Number analyzed (Participants) | 10 | 12 | 0
HCV RNA copies/mL plasma
  baseline | 7781148 (8662099) | 2320026 (3994266) |
  week 12 | 0 (0) | 0 (0) |
  week 24: number analyzed (Participants) | 9 | 11 | 0
  week 24 | 0 (0) | 0 (0) |

3. Secondary Outcome: Gene Expression Profiles
Description: Gene expression profiles in PBMC will be determined using RNA Seq
Time Frame: 24 weeks
Population: 9/10 Active injectors, 11/12 former injectors and 12/12 healthy volunteers completed the study. Healthy volunteers were only studied at baseline. No data for weeks 4, 12, 24.
Measure: Number; unit: RNA seq different from active IDU
Arm/Group | Active Injection Drug Use (IDU) | Former Injection Drug Use (Former IDU) | Healthy Volunteers
Number analyzed (Participants) | 9 | 11 | 12
RNA seq different from active IDU
  baseline | 9 | 11 | 12
  4 weeks: number analyzed (Participants) | 9 | 11 | 0
  4 weeks | 9 | 11 |
  12 weeks: number analyzed (Participants) | 9 | 11 | 0
  12 weeks | 9 | 11 |
  24 weeks: number analyzed (Participants) | 9 | 11 | 0
  24 weeks | 9 | 11 |

ADVERSE EVENTS:
Arm/Group | Active Injection Drug Use (IDU) | Former Injection Drug Use (Former IDU) | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Injection Drug Use (IDU) (N=10) | Former Injection Drug Use (Former IDU) (N=12) | Healthy Volunteers (N=12)
Drug overdose (General disorders) | 0 (0) | 1 (1) | 0 (0) — Study subject found dead. Autopsy consistent with multiple drug overdose. Likely cause of death cardiopulmonary arrest

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No